CLINICAL TRIAL: NCT01893879
Title: Placebo-Controlled Therapeutic Trial for the Prevention of Lymphedema in High Risk Patients
Brief Title: Placebo-Controlled Therapeutic Trial for the Prevention of Lymphedema
Acronym: PCTTPL
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: insufficient enrollment
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Stanley Rockson, Allan and Tina Neill Professor of Lymphatic Research and Medicine, Stanford University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: IRB-20651; BRSNSTU0028 (Other: OnCore); 4593 (Other: Stanford University Hospitals and Clinics)
Record Dates: First submitted 2013-07-02; First posted 2013-07-09 (Estimated); Results first posted 2017-05-18 (Actual); Last update posted 2017-05-18 (Actual); Status verified 2017-04

CONDITIONS: Lymphedema; Unspecified Adult Solid Tumor, Protocol Specific
MeSH Terms: conditions — Lymphedema | interventions — Drug Evaluation

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- (RS)2-(3-benzoylphenyl)-propionic acid (Experimental): Patients receive study drug PO TID for up to 1 year in the absence of disease progression or unacceptable toxicity.
  Laboratory biomarker analysis will be performed.
  Interventions: Drug: (RS)2-(3-benzoylphenyl)-propionic acid; Other: laboratory biomarker analysis
- placebo for study drug (Placebo Comparator): Patients receive placebo PO TID for up to 1 year in the absence of disease progression or unacceptable toxicity.
  Laboratory biomarker analysis will be performed.
  Interventions: Drug: placebo for study drug; Other: laboratory biomarker analysis

INTERVENTIONS:
Drug: placebo for study drug — Given PO
  Other Names: PLCB
  Arms: placebo for study drug
Drug: (RS)2-(3-benzoylphenyl)-propionic acid — Given PO
  Other Names: BPA
  Arms: (RS)2-(3-benzoylphenyl)-propionic acid
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
This randomized clinical trial studies an investigational drug in preventing lymphedema in patients at high risk after undergoing axillary lymph node dissection. The study drug may prevent lymphedema in patients undergoing axillary lymph node dissection.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate the efficacy of study drug in improving chronic lymphedema while further elucidating the role of inflammatory and lymphangiogenic processes in the pathogenesis of this disease.

OUTLINE: Patients are randomized to 1 of 2 treatment arms.

ARM I: Patients receive study drug orally (PO) thrice daily (TID) for up to 1 year in the absence of disease progression or unacceptable toxicity.

ARM II: Patients receive placebo PO TID for up to 1 year in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up for 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Axillary lymph node dissection within the preceding 12 months

Exclusion Criteria:

* Patients with active cancer
* Patients with lymphedema
* Infection or bleeding tendency
* Patients with medical contraindications to nonsteroidal anti-inflammatory drugs (NSAIDs), including history of allergies, know gastrointestinal intolerance
* Other serious systemic illness (e.g., renal failure, hepatic dysfunction, congestive heart failure, neurological or psychological impairment) that would impair the patients' ability to participate
* Persons not competent to consent
* Patients on aspirin therapy
* Minors (< 18 years of age)
* Pregnant and/or lactating women
* Males

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2014-04; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stanley Rockson, Principal Investigator — Stanford University Hospitals and Clinics
Locations (1):
- Stanford University Hospitals and Clinics, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Groups:
- (RS)2-(3-benzoylphenyl)-Propionic Acid: Patients receive study drug PO TID for up to 1 year in the absence of disease progression or unacceptable toxicity.
  Laboratory biomarker analysis will be performed.
  (RS)2-(3-benzoylphenyl)-propionic acid: Given PO
  laboratory biomarker analysis: Correlative studies
- Placebo for Study Drug: Patients receive placebo PO TID for up to 1 year in the absence of disease progression or unacceptable toxicity.
  Laboratory biomarker analysis will be performed.
  placebo for study drug: Given PO
  laboratory biomarker analysis: Correlative studies
Period: Overall Study
Arm/Group | (RS)2-(3-benzoylphenyl)-Propionic Acid | Placebo for Study Drug
Started | 7 | 7
Completed | 5 | 4
Not Completed | 2 | 3

BASELINE CHARACTERISTICS:
Groups:
- (RS)2-(3-benzoylphenyl)-Propionic Acid: Patients receive study drug three times daily, orally, for up to 1 year in the absence of disease progression or unacceptable toxicity.
  Laboratory biomarker analysis will be performed.
  (RS)2-(3-benzoylphenyl)-propionic acid: Given PO
  laboratory biomarker analysis: Correlative studies
- Placebo for Study Drug: Patients receive placebo three times daily, orally, for up to 1 year in the absence of disease progression or unacceptable toxicity.
  Laboratory biomarker analysis will be performed.
  placebo for study drug: Given PO
  laboratory biomarker analysis: Correlative studies
- Total: Total of all reporting groups
Arm/Group | (RS)2-(3-benzoylphenyl)-Propionic Acid | Placebo for Study Drug | Total
Number analyzed (Participants) | 7 | 7 | 14
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.8 (6.0) | 45.5 (10.1) | 45.2 (8.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 7 | 14
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 7 | 7 | 14

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Incidence of Lymphedema
Description: Participants were evaluated every 3 months up to one year post lymph node dissection
Time Frame: Up to 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | (RS)2-(3-benzoylphenyl)-Propionic Acid | Placebo for Study Drug
Number analyzed (Participants) | 5 | 4
Participants | 2 | 1

ADVERSE EVENTS:
Time Frame: Enrollment to 1 year post axillary lymph node dissection.
Arm/Group | (RS)2-(3-benzoylphenyl)-Propionic Acid | Placebo for Study Drug
Serious Adverse Events (participants affected / at risk) | 0/7 | 0/7
Other Adverse Events (participants affected / at risk) | 1/7 | 1/7
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | (RS)2-(3-benzoylphenyl)-Propionic Acid (N=7) | Placebo for Study Drug (N=7)
Swollen thumb (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) — 2 days of mild abdominal pain, resolved spontaneously

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No